CLINICAL TRIAL: NCT00445887
Title: Phase II Double Blind Randomized Trial Evaluating the Biologic Effect of Levonorgestrel on the Double Blind Randomized Trial Evaluating the Biologic Effect of Levonorgestrel on the Ovarian Epithelium in Women at High Risk for Ovarian Cancer
Brief Title: Levonorgestrel in Preventing Ovarian Cancer in Patients at High Risk for Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GOG-0214; NCI-2009-00588 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10-01367; CDR0000532268; GOG-0214; GOG-0214 (Other: Gynecologic Oncology Group); GOG-0214 (Other: DCP); GOG-0214 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2018-01-11 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Levonorgestrel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (levonorgestrel) (Experimental): Patients receive oral levonorgestrel once daily.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Levonorgestrel
- Arm II (placebo) (Placebo Comparator): Patients receive oral placebo once daily.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Levonorgestrel; Other: Placebo

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Levonorgestrel — Given orally
  Other Names: 18-Methylnorethisterone; D-(-)-Norgestrel; L-norgestrel; Mirena; Norplant; Plan B
Other: Placebo — Given orally
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase II trial is studying how well levonorgestrel works in preventing ovarian cancer in patients at high risk for ovarian cancer. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of levonorgestrel may prevent ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the impact of levonorgestrel on the relative frequency of apoptosis in the ovarian epithelium of patients at high risk for ovarian cancer.

SECONDARY OBJECTIVES:

I. Estimate the impact of this drug on proliferation and transforming growth factor-beta (TGF-beta) expression in the ovarian epithelium of these patients.

II. Assess the safety of this drug in these patients.

OUTLINE: This is a prospective, randomized, placebo-controlled, double-blind study. Patients are stratified according to menopausal status (premenopausal vs postmenopausal). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral levonorgestrel once daily.

ARM II: Patients receive oral placebo once daily.

In both arms, treatment continues for 4-6 weeks in the absence of disease progression or unacceptable toxicity, including on the day of surgery. Patients then undergo prophylactic salpingo-oophorectomy. After completion of study therapy, patients are followed at 1 year.

NOTE: * Patients who are unable to have surgery completed during the expected 4-6 weeks, may continue levonorgestrel or placebo for a time period no > 5 months. Patients unable to undergo surgery within 5 months are removed from the study.

ELIGIBILITY:
Inclusion Criteria:

* At increased genetic risk for ovarian cancer AND planning to undergo risk-reducing salpingo-oophorectomy (RRSO)

  * Has ≥ 1 intact ovary
* Patients enrolled on clinical trial GOG-0199 and planning to undergo RRSO allowed
* Submission of fixed ovarian tissue (FN01) required
* Must meet 1 of the following additional criteria:

  * Family of the patient has a documented deleterious BRCA1 or BRCA2 mutation and either the patient herself has tested positive for a deleterious BRCA1 or BRCA2 mutation or the patient has a first- or second-degree relative with a deleterious BRCA1 or BRCA2 mutation

    * No patient with a deleterious BRCA1 or BRCA2 mutation whose first- or second-degree relative has tested negative for the exact same mutation
  * The family contains members with ≥ 2 ovarian* and/or breast cancers among the first- or second-degree relatives (male relatives must be counted) of the patient within the same lineage (this condition may be satisfied by multiple primary cancers in the same person or, where breast cancer is required to meet this criterion, ≥ 1 breast cancer must have been diagnosed prior to menopause or at age ≤ 50 years if age at menopause is unknown)
  * The patient is of Ashkenazi Jewish ethnicity (lineage via the mother) with one first- degree or two second-degree maternal relatives with breast and/or ovarian cancer* (where breast cancer is required to meet this criterion, ≥ 1 breast cancer must have been diagnosed prior to menopause or at age ≤ 50 years if age at menopause is unknown)
  * The probability of carrying a BRCA1 or BRCA2 mutation, given the family pedigree of breast and ovarian cancers, exceeds 20%, as calculated by BRCAPRO
* No prior history of ovarian cancer, including low malignant potential cancers, or primary papillary serous carcinoma of the peritoneum
* No prior or concurrent history of breast cancer, including ductal carcinoma in situ (DCIS) of the breast

  * Women with a history of hormone receptor-negative breast cancer (both estrogen receptor-negative and progesterone receptor-negative) are eligible
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception prior to the prophylactic salpingo-oophorectomy
* No prior history of deep vein thrombosis, stroke, liver disease, or heart attack
* No prior history of myocardial infarction
* No known bleeding disorders or hypercoagulable states
* No other malignancy, including ductal carcinoma in situ, within 1 year of systemic therapy, except for nonmelanoma skin cancer
* No prior chemotherapy regimen lasting ≥ 12 months
* No oral or intrauterine hormonal contraception or hormonal replacement therapy within the past 3 months or injectable medroxyprogesterone within the past 12 months
* No intraperitoneal surgery within the past 3 months (including laparoscopy)
* No prior or concurrent radiotherapy to the pelvis
* No concurrent hormonal contraception
* No concurrent tamoxifen, raloxifene, estrogen, progesterone-like hormones, or other hormonal medication (including hormone replacement therapy)

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03-10 (Actual); Primary Completion 2013-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo C Rodriguez, Principal Investigator — Gynecologic Oncology Group
Locations (66):
- United States (66):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California San Diego, San Diego, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - Memorial Health University Medical Center, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol opened to accrual 03/10/2008 and closed 11/26/2012Women who were are at increased risk for ovarian cancer and were intending to undergo prophylactic salpingo-oopherectomy were randomized to Levenorgestrel (0.15 mg/day) or Placebo for 4 to 6 weeks.
Groups:
- Arm I (Levenorgestrel): Levenorgestrel (0.15 mg/day) for 4 to 6 weeks for 4 to 6 weeks
- Arm II (Placebo): Placebo for 4 to 6 weeks
Period: Overall Study
Arm/Group | Arm I (Levenorgestrel) | Arm II (Placebo)
Started | 33 | 31
Completed | 33 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Levenorgestrel) | Arm II (Placebo) | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0 | 0 | 0
  30-39 years | 4 | 6 | 10
  40-49 years | 14 | 13 | 27
  50-59 years | 14 | 9 | 23
  60-69 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Median Proportion Cells That Are Apoptotic in Epithelial Ovarian Tissue
Description: The median proportion of cells that are considered to be apoptotic are counted in the ovarian tissue sample, among the total number of cells available in the sample slide.
Time Frame: Surgical specimen (4 - 6 weeks after entry)
Population: Patients with evaluable slides. 14 of the cases did not have ovarian tissue available for evaluation. 50 cases were available for the primary analysis.
Measure: Median (Inter-Quartile Range); unit: proportion of total cells
Arm/Group | Arm I (Levenorgestrel) | Arm II (Placebo)
Number analyzed (Participants) | 26 | 24
proportion of total cells | .093 [.024 to .25] | .115 [.033 to .329]

2. Primary Outcome: Number of Participants With Adverse Events According to Grade as Determined by NCI CTCAE v.3.0
Description: Participants were graded using CTCAE v.30 criteria. Grade 1 is the least severe grade. Each adverse event lists criteria for grading, grade 1 being mild, up to grade 5. Grade 4 is generally life threatening. Grade 5 is death.
Time Frame: Up to 20 weeks
Population: All eligible and treated patients who had toxicity on study.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 1 CTCAE v 3.0 Arm I (Levonorgestrel): Number of patients on arm 1 who experienced a grade 1 event using CTCAE v 3.0
- Grade 2 CTCAE v 3.0 Arm 1 (Levonorgestrel): Number of patients on arm 1 who experienced a grade 2 event using CTCAE v 3.0
- Grade 3 CTCAE v 3.0 Arm 1 (Levonorgestrel): Number of patients on arm 1 who experienced a grade 3 event using CTCAE v 3.0
- Grade 4 CTCAE v3.0 Arm 1 Levonorgestrel): Number of patients on arm ! who experienced a grade 4 event using CTCAE v. 3.0
- Grade 5 CTCAE v3.0 Arm I (Levonorgestrel): Number of patients on arm I who experienced a grade 5 event using CTCAE v. 3.0
- Grade 1 CTCAE 3.0 Arm II (Placebo): Number of patients on arm II who experienced a grade 1 event using CTCAE v.30
- Grade 2 CTCAE 3.0 Arm II (Placebo): Number of patients on arm II who experienced a grade 2 event using CTCAE 3.0
- Grade 3 CTCAE 3.0 Arm II (Placebo): Number of patients on arm II who experienced a grade 3 event using CTCAE 3.0
- Grade 4 CTCAE 3.0 Arm II (Placebo): Number of patients on arm II who experienced a grade 4 event using CTCAE 3.0
- Grade 5 CTCAE 3.0 Arm II (Placebo): Number of patients on arm II who experienced a grade 5 event using CTCAE 3.0
Arm/Group | Grade 1 CTCAE v 3.0 Arm I (Levonorgestrel) | Grade 2 CTCAE v 3.0 Arm 1 (Levonorgestrel) | Grade 3 CTCAE v 3.0 Arm 1 (Levonorgestrel) | Grade 4 CTCAE v3.0 Arm 1 Levonorgestrel) | Grade 5 CTCAE v3.0 Arm I (Levonorgestrel) | Grade 1 CTCAE 3.0 Arm II (Placebo) | Grade 2 CTCAE 3.0 Arm II (Placebo) | Grade 3 CTCAE 3.0 Arm II (Placebo) | Grade 4 CTCAE 3.0 Arm II (Placebo) | Grade 5 CTCAE 3.0 Arm II (Placebo)
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 31 | 31 | 31 | 31 | 31
Participants
  Allergy/Immunology | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Constitutional Symptoms | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Cardiac | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dermatology/Skin | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Endocrine | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Gastrointestinal | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Renal/Genitourinary | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemorrhage/Bleeding | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Blood/Bone Marrow | 5 | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
  Infection | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Metabolic/Laboratory | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Neurology | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Pulmonary/Upper Respiratory | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain | 3 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
  Sexual/Reproductive Function | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

3. Secondary Outcome: Proportion of Proliferation as Measured by Ki-67
Time Frame: Time of surgery (4 to 6 weeks after entry)
Population: All eligible, treated patients with an evaluable sample.
Measure: Median (Inter-Quartile Range); unit: Proportion of cells exhibiting Ki-67
Arm/Group | Arm I (Levenorgestrel) | Arm II (Placebo)
Number analyzed (Participants) | 32 | 30
Proportion of cells exhibiting Ki-67 | .003 [0 to .008] | .008 [.002 to .028]

4. Secondary Outcome: Patients With High Expression of Transforming Growth Factor-beta 1
Time Frame: Baseline to time of surgery (4 to 6 weeks)
Population: All eligible, treated and evaluable for Transforming Growth factor-beta
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Levenorgestrel) | Arm II (Placebo)
Number analyzed (Participants) | 29 | 20
Participants | 6 | 3

5. Other Pre Specified Outcome: Median Proportion Cells That Are Apoptotic in Fallopian Tube Tissue
Description: The median proportion of cells that are considered to be apoptotic are counted in the fallopian tube tissue sample, among the total number of cells available in the sample slide
Time Frame: Surgical specimen (4-6 weeks after entry)
Population: Patients with evaluable slides
Measure: Median (Inter-Quartile Range); unit: proportion of total cells
Arm/Group | Arm I (Levenorgestrel) | Arm II (Placebo)
Number analyzed (Participants) | 32 | 30
proportion of total cells | .205 [.07 to .395] | .079 [.01 to .25]

ADVERSE EVENTS:
Time Frame: Study Treatment - 4 - 6 weeks from enrollment
Arm/Group | Arm I (Levenorgestrel) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 16/33 | 14/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Levenorgestrel) (N=33) | Arm II (Placebo) (N=31)
Allergy/Immunology - Other (Immune system disorders) | 1 | 0
Rhinitis (Immune system disorders) | 0 | 1
Neutrophils (Blood and lymphatic system disorders) | 1 | 0
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 0 | 1
Leukocytes (Blood and lymphatic system disorders) | 0 | 2
Hemoglobin (Blood and lymphatic system disorders) | 6 | 3
Hypertension (Cardiac disorders) | 1 | 0
Sweating (General disorders) | 1 | 0
Fever (General disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 0 | 1
Hot Flashes (Endocrine disorders) | 1 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Distention (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Hemorrhage, Gu - Vagina (Vascular disorders) | 3 | 1
Infection - Other (Infections and infestations) | 1 | 0
Inf Unknown Anc: Bronchus (Infections and infestations) | 0 | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 1 | 0
Inf Unknown Anc: Colon (Infections and infestations) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Pain: Chest /Thorax Nos (General disorders) | 1 | 0
Pain: Head/Headache (General disorders) | 2 | 2
Pain: Back (General disorders) | 0 | 1
Pain: Bladder (General disorders) | 1 | 0
Pain: Abdominal Pain Nos (General disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Frequency (Renal and urinary disorders) | 1 | 0
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 1 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No